CLINICAL TRIAL: NCT01725165
Title: A Randomized Phase II Study Assessing the Efficacy of Local Consolidative Therapy for Non-Small Cell Lung Cancer Patients With Induced Oligometastatic Disease
Brief Title: Surgery and/or Radiation Therapy or Standard Therapy and/or Clinical Observation in Treating Patients With Previously Treated Stage IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0618; NCI-2012-02874 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0618 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Recurrent Lung Non-Small Cell Carcinoma; Stage IV Non-Small Cell Lung Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Watchful Waiting; Observation

ARMS (2):
- Arm I (immediate LCT) (Experimental): Patients undergo ablation of all residual local and metastatic sites of disease by surgery and/or EBRT. After completion of LCT, patients undergo either surveillance or maintenance treatment at the discretion of the treating physician.
  Interventions: Radiation: External Beam Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Procedure: Therapeutic Conventional Surgery
- Arm II (delayed/no LCT) (Active Comparator): Patients undergo standard maintenance therapy or clinical observation, based on physician choice. Patients may cross-over to Arm I due to RECIST progression or toxicity at the treating physician's discretion.
  Interventions: Other: Clinical Observation; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Procedure: Standard Follow-Up Care

INTERVENTIONS:
Other: Clinical Observation — Undergo clinical observation
  Other Names: observation
  Arms: Arm II (delayed/no LCT)
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation
  Arms: Arm I (immediate LCT)
Other: Laboratory Biomarker Analysis — Optional correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Standard Follow-Up Care — Undergo standard maintenance therapy
  Arms: Arm II (delayed/no LCT)
Procedure: Therapeutic Conventional Surgery — Undergo surgery
  Arms: Arm I (immediate LCT)

SUMMARY:
This randomized phase II trial studies how well surgery and/or radiation therapy or standard therapy and/or clinical observation works in treating patients with previously treated stage IV non-small cell lung cancer. Radiation therapy uses high energy x-rays to kill tumor cells. Giving surgery and/or radiation therapy may be more effective than standard therapy and/or clinical observation in patients with previously treated non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether oligometastatic non-small cell lung cancer (NSCLC) patients with no disease progression after first line therapy have prolonged progression free survival (PFS) when treated with local consolidation therapy (LCT) of residual disease (radiation or surgery) followed by maintenance or surveillance as per physician choice compared with no LCT.

SECONDARY OBJECTIVES:

I. Determine the overall survival. II. Safety/tolerability of LCT. III. Time to progression of prior metastatic lesions. IV. Time to appearance of new metastases (central nervous system [CNS] vs. extra-CNS, treated lesion vs. new site).

V. Quality of life (QOL).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I (IMMEDIATE LCT): Patients undergo ablation of all residual local and metastatic sites of disease by surgery and/or external beam radiation therapy (EBRT). After completion of LCT, patients undergo either surveillance or maintenance treatment at the discretion of the treating physician.

ARM II (DELAYED/NO LCT): Patients undergo standard maintenance therapy or clinical observation, based on physician choice. Patients may cross-over to Arm I due to Response Evaluation Criteria in Solid Tumors (RECIST) progression or toxicity at the treating physician's discretion.

After completion of study treatment, patients are followed up for 9 months.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 ENROLLMENT: the patient has a diagnosis of pathologically confirmed NSCLC by tumor biopsy and/or fine-needle aspiration; mixed tumors will be categorized by the predominant cell type
* STEP 1 ENROLLMENT: the patient has a diagnosis of American Joint Committee on Cancer (AJCC) 7th Edition stage IV NSCLC
* STEP 1 ENROLLMENT: three or less metastatic lesions (not sites); each lesion (including a satellite nodule) will individually be counted as one, and intrathoracic lymph node involvement (defined here as hilar, mediastinal, or supraclavicular nodes, N1-N3) will collectively be counted as one; in addition, patients can receive treatment to CNS lesions or other symptomatic lesions requiring urgent local therapy prior to randomization, but these lesions will be counted towards the total number after chemotherapy, and patients will only be eligible if there are remaining sites amenable to local therapy after up-front systemic therapy
* STEP 1 ENROLLMENT: standard induction chemotherapy planned defined as: at least 4 cycles of platinum doublet chemotherapy for metastatic disease (with or without bevacizumab); if the patient is known to be EGFR mutation positive, erlotinib, afatinib, or gefitinib for >= 3 months, or for patients with known EML4-ALK fusions, crizotinib for >= 3 months
* STEP 2 ENROLLMENT AND RANDOMIZATION: the patient has a diagnosis of pathologically confirmed NSCLC by tumor biopsy and/or fine-needle aspiration; mixed tumors will be categorized by the predominant cell type
* STEP 2 ENROLLMENT AND RANDOMIZATION: the patient has a diagnosis of American Joint Committee on Cancer (AJCC) 7th edition stage IV NSCLC
* STEP 2 ENROLLMENT AND RANDOMIZATION: completion of standard induction chemotherapy planned defined as: at least 4 cycles of platinum doublet chemotherapy for metastatic disease (with or without bevacizumab); if the patient is known to be EGFR mutation positive, erlotinib, afatinib, or gefitinib for >= 3 months, or for patients with known EML4-ALK fusions, crizotinib; note that it is not mandatory to check EGFR mutation or EML4-ALK status prior to entry, but patients that receive options 2 or 3 should have had these molecular tests performed
* STEP 2 ENROLLMENT AND RANDOMIZATION: less than or equal to three metastatic lesions and no evidence of disease progression based on RECIST criteria; note that patients that had > 3 metastatic lesions in Step 1 may be eligible for enrollment in Step 2 if the number of metastatic sites is reduced to three or less
* STEP 2 ENROLLMENT AND RANDOMIZATION: the patient's Eastern Cooperative Oncology Group (ECOG) performance status is =< 2 at study entry
* STEP 2 ENROLLMENT AND RANDOMIZATION: absolute neutrophil count (ANC) >= 1,500/mm^3 within 3 weeks of study entry
* STEP 2 ENROLLMENT AND RANDOMIZATION: platelet count >= 100,000/mm^3 within 3 weeks of study entry
* STEP 2 ENROLLMENT AND RANDOMIZATION: white blood cells (WBC) >= 3,000/mm^3 within 3 weeks of study entry
* STEP 2 ENROLLMENT AND RANDOMIZATION: hemoglobin >= 9 g/dL within 3 weeks of study entry
* STEP 2 ENROLLMENT AND RANDOMIZATION: the patient must be a suitable candidate for LCT (radiotherapy and/or surgery) to every site of disease, as determined by the treating physician(s); consultation with a multidisciplinary team, including a medical oncologist, radiation oncologist, and thoracic surgeon, is encouraged but not required
* STEP 2 ENROLLMENT AND RANDOMIZATION: concurrent chemoradiation is permitted as consolidative therapy; the following concurrent therapies are permitted: tyrosine kinase inhibitors (i.e. erlotinib) - can be delivered with both hypofractionated (>= 3 Gray [Gy] per fraction) and standard fractionated radiation therapy (< 3 Gy per fraction); platinum-based chemotherapy - standard fractionated radiation therapy (< 3 Gy per fraction)
* STEP 2 ENROLLMENT AND RANDOMIZATION: bevacizumab will not be permitted within 2 weeks of the initiation of the radiation therapy course
* STEP 2 ENROLLMENT AND RANDOMIZATION: treatment to central nervous system lesions, such as the brain or spine (prior to first line systemic therapy), or symptomatic lesions requiring urgent palliative radiation, is permitted prior to randomization, in which case the patient would be randomized to treatment of other metastatic sites or the primary sites (based on the disease remaining after first-line treatment); these treated lesions should be counted towards the total number of metastases at the time of enrollment
* STEP 2 ENROLLMENT AND RANDOMIZATION: the patient has signed informed consent
* STEP 2 ENROLLMENT AND RANDOMIZATION: women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation and for six (6) months after discontinuation of the study drugs; childbearing potential will be defined as women who have had menses within the past 12 months, who have not had tubal ligation, hysterectomy or bilateral oophorectomy; should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately; the patient, if a man, agrees to use effective contraception or abstinence for the duration of study participation and for six (6) months after discontinuation of the study drugs

Exclusion Criteria:

* STEPS 1 AND 2 AND RANDOMIZATION
* The patient has a history of uncontrolled angina, arrhythmias, or congestive heart failure
* Patients with a history of malignant pleural effusions are not eligible; pleural effusions considered by the investigator too small for a diagnostic thoracentesis are permissible
* Patient is pregnant (confirmed by serum beta- b-human chorionic gonadotropin [HCG] if applicable) or is breastfeeding
* Presence of significant third space fluid which cannot be controlled by drainage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-11-28 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Tang, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (2):
  - University of Colorado, Denver, Colorado
  - M D Anderson Cancer Center, Houston, Texas
- London Health Sciences Centre-South Street, London, Ontario, Canada

REFERENCES:
- [Derived] Tang C, Lee WC, Reuben A, Chang L, Tran H, Little L, Gumbs C, Wargo J, Futreal A, Liao Z, Xia X, Yi X, Swisher SG, Heymach JV, Gomez D, Zhang J. Immune and Circulating Tumor DNA Profiling After Radiation Treatment for Oligometastatic Non-Small Cell Lung Cancer: Translational Correlatives from a Mature Randomized Phase II Trial. Int J Radiat Oncol Biol Phys. 2020 Feb 1;106(2):349-357. doi: 10.1016/j.ijrobp.2019.10.038. Epub 2019 Oct 31. PMID 31678224
- [Derived] Gomez DR, Blumenschein GR Jr, Lee JJ, Hernandez M, Ye R, Camidge DR, Doebele RC, Skoulidis F, Gaspar LE, Gibbons DL, Karam JA, Kavanagh BD, Tang C, Komaki R, Louie AV, Palma DA, Tsao AS, Sepesi B, William WN, Zhang J, Shi Q, Wang XS, Swisher SG, Heymach JV. Local consolidative therapy versus maintenance therapy or observation for patients with oligometastatic non-small-cell lung cancer without progression after first-line systemic therapy: a multicentre, randomised, controlled, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1672-1682. doi: 10.1016/S1470-2045(16)30532-0. Epub 2016 Oct 24. PMID 27789196
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: 11/28/2012 to 02/01/2016 ; Location: Multi-center trial that recruited patients at three different hospital sites (MD Anderson Cancer Center, Houston, TX; London Health Sciences Center, London, Ontario; and The University of Colorado, Aurora, CO) 9 patients in the MT/O group received LCT after progression. The remaining 15 did not.
Pre-assignment Details: Three patients in the MT/O arm who crossed over to receive LCT before progression were excluded because they did not adhere to either arm of the study.
Groups:
- LCT Arm: LCT with radiation therapy or surgery followed by standard maintenance or observation
- MT/O Arm: Standard maintenance (chosen by the treating physician from predefined set of standard of care options) or observation
Period: Overall Study
Arm/Group | LCT Arm | MT/O Arm
Started | 25 | 24
Completed | 14 | 6
Not Completed | 11 | 18
Not completed — Death | 11 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCT Arm | MT/O Arm | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 11 | 10 | 21
Age, Continuous [Median (Full Range); unit: Years] | 63 [43 to 83] | 61 [43 to 80] | 61 [43 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 12 | 10 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 20 | 18 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 49
Patient Characteristics [Number; unit: participants] — Age (years), Sex, Ethnicity, Tumor histology, Timing of metastatic disease, Number of of nonregional metastases after initial systemic therapy, Response to first-line chemotherapy, CNS metastases, Nodal status, Mutation type
  participants | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: The measurement of overall survival of patients from the start of trial participation until the time their disease progresses or death of the patient. The outcome measures were stratified per the randomization on protocol. The results were not reclassified based on later sequencing. This was all done in accordance to the protocol document.
Time Frame: 16.6 months to 41.2 months for all patients in both LCT and MT/O group
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LCT Arm | MT/O Arm
Number analyzed (Participants) | 25 | 24
Months | 14.2 [7.4 to 23.1] | 4.4 [2.2 to 8.3]

2. Secondary Outcome: Time to New Lesion Progression
Description: The measurement of time to new lesion progression of patients from the start of trial participation until the time their disease progresses. The outcome measures were stratified per the randomization on protocol. The results were not reclassified based on later sequencing. This was all done in accordance to the protocol document.
Time Frame: 5.7 to 24.3 months (LCT group); 4.4 to 8.3 months (MT/O group)
Measure: Median (Full Range); unit: Months
Arm/Group | LCT Arm | MT/O Arm
Number analyzed (Participants) | 25 | 24
Months | 14.2 [5.7 to 24.3] | 6 [4.4 to 8.3]

ADVERSE EVENTS:
Time Frame: From baseline to 61.4 months post treatment.
Description: At the time of cross over they came off active study follow up. No adverse events were assessed after cross over.
Arm/Group | LCT Arm | MT/O Arm
All-Cause Mortality (participants affected / at risk) | 11/25 | 18/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 14/25 | 12/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCT Arm (N=25) | MT/O Arm (N=24)
Fatigue (General disorders) | 1 | 1
Renal Insufficiency (Renal and urinary disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Esophagitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1
Odynophagia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Peripheral Sensory Neuropathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Neuropathy (Nervous system disorders) | 1 | 1
Peripheral Neuropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysphagia (General disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1
Fever (General disorders) | 0 | 1
Hoarseness (General disorders) | 0 | 1
Pain (of neck) (General disorders) | 1 | 0
Pain (of chestwall) (General disorders) | 1 | 0
Watery eyes (General disorders) | 0 | 1
Back Pain (General disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Short of Breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diverticulitis (Gastrointestinal disorders) | 1 | 0
Chronic Renal Failure (Renal and urinary disorders) | 0 | 1
Blurred Vision (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Depression (General disorders) | 0 | 1
Anion Gap Decrease (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Left rib pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cellulitis (General disorders) | 0 | 1
Thrush (Infections and infestations) | 1 | 0
Abdominal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Anorexia (General disorders) | 1 | 0
Edema (Blood and lymphatic system disorders) | 1 | 0
Dry Eyes (General disorders) | 1 | 0
Hypoxemia (Blood and lymphatic system disorders) | 1 | 0
Hyperkalemia (Blood and lymphatic system disorders) | 1 | 0
Mucositis Oral (Skin and subcutaneous tissue disorders) | 0 | 1
Insomnia (General disorders) | 1 | 0
Headache (General disorders) | 1 | 1
Urinary difficulties (Renal and urinary disorders) | 0 | 0
Weight loss (General disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Cough (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT01725165/Prot_SAP_000.pdf